CLINICAL TRIAL: NCT05806177
Title: Safety, Tolerability and Pharmacokinetics of AD16 Tablets After Multiple Administration in Healthy Chinese Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of AD16 Tablets After MAD in Healthy Chinese Adult Subjects
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South China Center For Innovative Pharmaceuticals (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCCIP-AD16-2018-03
Record Dates: First submitted 2023-03-01; First posted 2023-04-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, placebo-controlled, double-blind, dose-increasing study design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD16 (Experimental): AD16 tablets should be administered only in the morning on the day of the first dose and on the ninth day after the first dose. Fasting is required for at least 10 h before administration.Two dosing cohorts received AD16 From the third day to the eighth day, the medicine was administered twice a day, 1 h before breakfast, 1 h before dinner or 2 h after dinner, with a 12 h interval (time window ±1 h).The duration of oral AD16 tablets was nine days.
  Interventions: Drug: AD16 30mg、40mg
- AD16 placebo (Placebo Comparator): AD16 placebo tablets should be administered only in the morning on the day of the first dose and on the ninth day after the first dose. Fasting is required for at least 10 h before administration.Two dosing cohorts received AD16 placebo From the third day to the eighth day, the medicine was administered twice a day, 1 h before breakfast, 1 h before dinner or 2 h after dinner, with a 12 h interval (time window ±1 h).The duration of oral AD16 placebo tablets was nine days.
  Interventions: Drug: AD16 Placebo 30mg、40mg

INTERVENTIONS:
Drug: AD16 30mg、40mg — AD16 was taken continuously.Firstly, a 30 mg (bid) multiple dose study was conducted, followed by a 40 mg (bid) multiple dose study
  Arms: AD16
Drug: AD16 Placebo 30mg、40mg — AD16 placebo was taken continuously.Firstly, a 30 mg (bid) multiple dose study was conducted, followed by a 40 mg (bid) multiple dose study
  Arms: AD16 placebo

SUMMARY:
This single-center, randomized, placebo-controlled, double-blind, dose-increasing study was designed to evaluate the safety, tolerability, and pharmacokinetics of multiple successive dosing in healthy Chinese adult subjects.In this study, 20 healthy adult subjects were enrolled in a multi-dose study in the 30mg and 40mg groups.

DETAILED DESCRIPTION:
In this study, subjects were given multiple doses in the corresponding dose group

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects were aged 18-45 years (including boundary values), male and female.
2. Weight ≥50kg (male) or ≥45kg (female), and body mass index (BMI) of 19-24kg/m2 (including the boundary values at both ends).
3. Have fully understood this study, voluntarily participated in it, and signed the Informed Consent.
4. Subjects are able to communicate well with researchers and complete the study according to protocol.
5. The subjects were deemed to be in good health based on physical examination, medical history, vital signs, electrocardiogram, chest X-ray, abdominal ultrasound, and laboratory tests.
6. Subject (including partner) is willing to have no pregnancy plan for the next 30 days (female subject) or 90 days (male subject) and is willing to use effective contraception.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or HIV antibody.
2. The patient has symptoms or related history of any serious disease, including but not limited to heart, liver, kidney, or other acute or chronic digestive tract or respiratory tract diseases, as well as diseases of the blood, endocrine, neurological, psychiatric and other systems, or any other disease or physiological condition that can interfere with the study results.
3. A history of postural hypotension with frequent episodes.
4. A history of frequent nausea or vomiting due to any cause.
5. Any clear history of drug or food allergies, especially allergies to ingredients similar to the drugs in this study.
6. Have special dietary requirements and cannot comply with the uniform diet provided by the clinical research center.
7. Previous drug abuse history or positive urine drug screening during screening period.
8. Smokers who smoked more than 5 cigarettes a day in the 3 months before the test.
9. Heavy drinkers or regular drinkers in the 6 months prior to the study screening, who drank more than 14 units of alcohol per week (1 unit of alcohol ≈360 mL beer or 45 mL 40% spirits or 150 mL wine) or had a positive alcohol breath test during the screening period.
10. Excessive consumption of tea, coffee (more than 6 cups) and/or caffeinated beverages (more than 1L) per day.
11. Take food or drink rich in xanthine, grapefruit or alcohol, caffeine (e.g., dragon fruit, mango, grapefruit, chocolate, coffee or tea) within 48 hours before administration.
12. Surgical procedures, transfusions of blood or blood components in the month prior to study screening.
13. Blood loss or donation of more than 400 mL in the 2 months prior to screening.
14. Participated in other clinical studies and took experimental drugs within 3 months prior to study screening.
15. Study participants who had received any medication in the 28 days prior to screening.
16. Pregnant or lactating women or women who have had unprotected sex within 14 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | day-7 to day11
  The number of adverse events
Serious adverse events | day-7 to day11
  The number of serious adverse events
Number of participants with abnormal laboratory test results | Screening period (day-7 to day-2) and day11
  Laboratory tests include Blood routine, blood biochemistry, coagulation function and urine routine, etc.
Number of participants with abnormal vital signs | Screening period（day-7 to day-1）、days1、4、5、6、8、9
  Pulse, blood pressure, body temperature and respiratory rate were observed at different time points before and after medication.
Number of participants with abnormal 12-lead electrocardiogram readings | Screening period（day-7 to day-2）、days1、6、11
  Abnormal12-lead electrocardiogram
Number of participants with abnormal physical examination findings | Screening period（day-7 to day-2）、days11
  The skin, mucosa, lymph nodes, head, neck, chest, abdomen, spine/limbs and nervous system were observed at different time points before and after medication.
Concomitant medication | Up to day 11
  Any concomitant medication

SECONDARY OUTCOMES:
Tmax of AD16 | Up to day 11
  Time to reach the maximum (peak) plasma concentration following drug administration
Cmax of AD16 | Up to day 11
  Maximum (peak) plasma drug concentration
t1/2z of AD16 | Up to day 11
  Elimination half-life (to be used in a one-compartment or noncompartmental model)
AUC 0-∞ of AD16 | Up to day 11
  Area under the plasma concentration-time curve（AUC） from time zero to infinity
AUC 0-t of AD16 | Up to day 11
  Area under the plasma concentration-time curve（AUC） from time zero to time t
Vd/F of AD16 | Up to day 11
  Apparent volume of distribution after non-intravenous administration
CL/F of AD16 | Up to day 11
  CL/F is defined as the ratio of total clearance(CL) to bioavailability(F).
λz of AD16 | Up to day 11
  Terminal disposition rate constant/terminal rate constant
AUC 0-48h of AD16 | Up to day 11
  Area under the plasma concentration-time curve from time zero to time 48h
AUC_%Extrap of AD16 | Up to day 11
  AUC_%Extrap is residual area percentage
Tmax,ss of AD16 | Up to day 11
  Time to reach the maximum (peak) plasma concentration following drug administration at steady state
Cmax, ss of AD16 | Up to day 11
  Maximum (peak) steady-state plasma drug concentration during a dosage interval
Cavg,ss of AD16 | Up to day 11
  Cavg,ss is the steady-state mean concentration
t1/2,ss of AD16 | Up to day 11
  Elimination half-life（steady state ）
AUC 0-τ,ss of AD16 | Up to day 11
  The area under the plasma concentration-time curve during a dosing interval at steady state
AUC 0-48h,ss of AD16 | Up to day 11
  Area under the plasma concentration-time curve from the last dose to 48 h
AUC 0-∞,ss of AD16 | Up to day 11
  The area under the plasma concentration-time curve is extrapolated from the last dose to infinity
CL/F,ss of AD16 | Up to day 11
  CL/F is defined as the ratio of total clearance(CL) to bioavailability(F)（steady state ）
Rac of AD16 | Up to day 11
  Rac is accumulation ratio
DF of AD16 | Up to day 11
  Degree of fluctuation（DF）Percentage fluctuation in steady state = 100 × (Cmax,ss -Cmin,ss)/Cavg,ss
Vd/F,ss of AD16 | Up to day 11
  Apparent volume of distribution after non-intravenous administration （steady state ）

CONTACTS AND LOCATIONS:
Locations (1):
- The Central South University Xiang Ya Hospital, Changsha, China

REFERENCES:
- [Derived] Peng D, Xu S, Zou T, Wang Y, Ouyang W, Zhang Y, Dong C, Li D, Guo J, Shen Q, Hu X, Zhou W, Li X, Qin Q. Safety, tolerability, pharmacokinetics and effects of diet on AD16, a novel neuroinflammatory inhibitor for Alzheimer's disease: a randomized phase 1 study. BMC Med. 2023 Nov 23;21(1):459. doi: 10.1186/s12916-023-03126-9. PMID 37996817